CLINICAL TRIAL: NCT07379931
Title: Randomized Clinical Trial to Analyze the Efficacy of a Liquid Carob Extract on the Glucose Metabolism of Subjects With Prediabetes.
Brief Title: Evaluating a Liquid Extract of Carob to Improve Blood Sugar in People With Prediabetes
Acronym: GLIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Medical degree, San Antonio Technologies - San Antonio Catholic University of Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UCAMCFE-00037
Record Dates: First submitted 2025-12-17; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Prediabetes (Insulin Resistance, Impaired Glucose Tolerance)
Keywords: Prediabetes; Glucose; Carob; Placebo
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Glucose Intolerance | interventions — locust bean gum; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carob Liquid (Experimental): Nutritional product: liquid carob extract.
  Interventions: Dietary Supplement: Carob extract
- Control group (Placebo Comparator): Nutritional product: placebo
  Interventions: Dietary Supplement: Control product

INTERVENTIONS:
Dietary Supplement: Carob extract — Consumo durante 90 días. La dosis diaria del producto es de 6,66 g/día, dividida en dos dosis de 3,33 g/dosis al día. El producto debe tomarse 30 minutos antes de las dos comidas principales del día.
  Arms: Carob Liquid
Dietary Supplement: Control product — Identical characteristics to the product under study. Consumption for 90 days, twice a day.
  Arms: Control group

SUMMARY:
This study evaluates whether a liquid carob extract can improve blood glucose levels in individuals with prediabetes. Participants are selected according to predefined health criteria and randomly assigned to two groups: one group receives the carob extract and the other receives an inert liquid (placebo). Blood samples are collected and glucose-related parameters are measured throughout the study to assess changes over time. The objective is to determine whether this extract may contribute to better glycemic control and help prevent progression to diabetes.

DETAILED DESCRIPTION:
This study is designed to assess the efficacy of a carob extract on glucose metabolism in individuals presenting impaired fasting glucose or elevated glycated hemoglobin levels, without current antidiabetic pharmacological treatment. Participants will consume the extract for 90 days, and metabolic outcomes will be compared with baseline values.

Secondary objectives include assessing changes in glucose area under the curve and peak glucose levels following an oral glucose tolerance test; evaluating variations in fasting glucose and fasting insulin levels after 90 days of intake; and determining changes in peripheral insulin resistance using the HOMA-IR and QUICKI indices. Additionally, potential effects on body composition will be assessed in individuals with abnormal fasting glucose or HbA1c values. Product safety will be monitored and analyzed throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes aged between 18 and 65.
* Diagnosis of prediabetes according to the American Diabetes Association (at least one of the following criteria):
* Impaired fasting glucose (100-125 mg/dL)
* Glucose intolerance (oral glucose tolerance test with blood glucose between 140-199 mg/dL after 2 hours).
* Glycated hemoglobin between 5.7 and 6.4%
* Subjects with a body mass index between 20-35 kg/m2.
* Stable eating habits: no weight gain or loss of more than 5 kg in the last ten weeks.
* Volunteers capable of understanding the clinical study and willing to comply with the study procedures and requirements.

Exclusion Criteria:

* Use of medications that may interfere with glucose metabolism.
* Subjects with a history of any type of liver or kidney disease.
* Alcohol consumption greater than 20 g/day.
* History of allergic hypersensitivity or poor tolerance to any component of the products under study.
* Participation in another clinical trial in the three months prior to the study.
* Unwillingness or inability to comply with clinical trial procedures.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of blood glucose during the oral glucose tolerance test | This assessment will be performed at baseline, on day 45, and on day 90.
  The area under the curve (AUC) of blood glucose during an oral glucose tolerance test (OGTT) with a glucose load of 50 g will be calculated. Capillary blood glucose levels will be measured at 0, 15, 30, 45, 60, 90, and 120 minutes after glucose ingestion.
Glycosylated hemoglobin (HbA1c) | Measurements will be taken at baseline, on day 45, and on day 90.
  Fasting glycosylated hemoglobin (HbA1c) will be measured in venous blood samples to assess long-term glycemic control.

SECONDARY OUTCOMES:
Area under the curve (AUC) of blood insulin during the oral glucose tolerance test | This assessment will be performed at the start of the study, on day 45, and on day 90.
  The area under the curve (AUC) of insulinemia will be calculated during an oral glucose tolerance test (OGTT) with a glucose load of 50 g. Serum insulin levels will be measured at 0, 15, 30, 45, 60, 90, and 120 minutes after glucose ingestion.
Insulin resistance and insulin sensitivity indices | Both indices will be calculated at baseline, day 45, and day 90.
  Peripheral insulin resistance and insulin sensitivity will be assessed using validated surrogate indices derived from fasting glucose and insulin levels: HOMA-IR (Homeostasis Model Assessment of Insulin Resistance) QUICKI (Quantitative Insulin Sensitivity Quotient).
Body composition analysis | These measurements will be taken at the beginning, on day 45, and on day 90.
  Body composition will be assessed using bioelectrical impedance analysis (BIA), providing estimates of fat mass, lean mass, and total body water.
Liver safety variables | These measurements will be performed at baseline, on day 45, and on day 90.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)
Adverse events | At 12 weeks after consumption
  It will be evaluated at each of the visits.

CONTACTS AND LOCATIONS:
Overall Officials: Fco Javier López Roman, Medical degree, Principal Investigator — Catholic University of Murcia
Locations (1):
- UCAM HiTech, Sport & Health Innovation Hub, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No